CLINICAL TRIAL: NCT01779765
Title: The Efficacy of Hydrolyzed Guar Gum ( PHGG) in the Treatment of Patients With Irritable Bowel Syndrome- a Double Blind, Placebo - Controlled, Randomized Study
Brief Title: The Efficacy of Hydrolyzed Guar Gum ( PHGG) in the Treatment of Patients With Irritable Bowel Syndrome (IBS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-12-NV-242-CTIL
Record Dates: First submitted 2013-01-10; First posted 2013-01-30 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2013-01

CONDITIONS: IBS
Keywords: IBS; Diarrhea; Constipation; Fibers
MeSH Terms: conditions — Diarrhea; Constipation | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PHGG (Experimental): 2.5gr per day for the first week and then 5gr per day for 11 weeks.
  Interventions: Dietary Supplement: PHGG
- Maltodextrin (Placebo Comparator): 2.5gr per day for the first week and then 5gr per day for 11 weeks.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: PHGG
  Arms: PHGG
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
This study objective is to assess the short and long term effects of partially hydrolyzed guar gum (PHGG) administration on clinical symptoms of IBS and quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the Rome III criteria for IBS.
* Aged 20-68 years at the time of screening.
* Provision of written informed consent.
* Commitment of availability throughout the 6 months study period.

Exclusion Criteria:

* Major abdominal surgery in the past.
* The presence of any active (organic)GI disease.
* Past or present major medical or psychiatric illness.
* Any concomitant disease.
* Alarming symptoms (rectal bleeding, weight loss, etc.)
* Pregnancy.
* Family history of colorectal carcinoma or inflammatory bowel disease (IBD).
* Abnormal laboratory studies (blood biochemistry , liver enzymes,complete blood count), abnormal thyroid function.
* Non-adjusted diet in the case of lactose or gluten intolerance.
* Recent travel to regions with endemic parasitic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in IBS score. | 2 years
  IBS scoring - Francis severity IBS score.

SECONDARY OUTCOMES:
Quality questionnaire | 2 years
  Quality of life - by the IBS - quality of life questionnaire - Drossman Patrick.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Jones J, Boorman J, Cann P, Forbes A, Gomborone J, Heaton K, Hungin P, Kumar D, Libby G, Spiller R, Read N, Silk D, Whorwell P. British Society of Gastroenterology guidelines for the management of the irritable bowel syndrome. Gut. 2000 Nov;47 Suppl 2(Suppl 2):ii1-19. doi: 10.1136/gut.47.suppl_2.ii1. No abstract available. PMID 11053260
- [Background] Mertz HR. Irritable bowel syndrome. N Engl J Med. 2003 Nov 27;349(22):2136-46. doi: 10.1056/NEJMra035579. No abstract available. PMID 14645642
- [Background] Parisi GC, Zilli M, Miani MP, Carrara M, Bottona E, Verdianelli G, Battaglia G, Desideri S, Faedo A, Marzolino C, Tonon A, Ermani M, Leandro G. High-fiber diet supplementation in patients with irritable bowel syndrome (IBS): a multicenter, randomized, open trial comparison between wheat bran diet and partially hydrolyzed guar gum (PHGG). Dig Dis Sci. 2002 Aug;47(8):1697-704. doi: 10.1023/a:1016419906546. PMID 12184518
- [Derived] Niv E, Halak A, Tiommny E, Yanai H, Strul H, Naftali T, Vaisman N. Randomized clinical study: Partially hydrolyzed guar gum (PHGG) versus placebo in the treatment of patients with irritable bowel syndrome. Nutr Metab (Lond). 2016 Feb 6;13:10. doi: 10.1186/s12986-016-0070-5. eCollection 2016. PMID 26855665